CLINICAL TRIAL: NCT05297045
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Ranging Study of Oral RGT001-075 in Adult Patients With Uncontrollable Type 2 Diabetes Mellitus on Metformin Therapy
Brief Title: A Study of Oral GLP1RA RGT001-075 in Adults With Type 2 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to financial constraint.
Sponsor: Regor Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGT001-075_01-201
Record Dates: First submitted 2022-02-24; First posted 2022-03-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Group A (Experimental)
  Interventions: Drug: RGT001-075
- Dose Group B (Experimental)
  Interventions: Drug: RGT001-075
- Dose Group C (Experimental)
  Interventions: Drug: RGT001-075
- Dose Group D (Experimental)
  Interventions: Drug: RGT001-075
- Dose Group E (Experimental)
  Interventions: Drug: RGT001-075
- Dose Group F (Experimental)
  Interventions: Drug: RGT001-075
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RGT001-075 — Oral GLP1 Receptor Agonist
  Arms: Dose Group A; Dose Group B; Dose Group C; Dose Group D; Dose Group E; Dose Group F
Other: Placebo — Placebo comparator
  Arms: Placebo Group

SUMMARY:
This is a phase 2 study designed to evaluate the efficacy of daily (QD) oral RGT001-075 GLP1 receptor agonist relative to placebo after up to 16 weeks of double-blind treatment as determined by mean change from baseline in HbA1c in adult patients with Type 2 Diabetes Mellitus (T2DM) who have inadequate glycemic control with diet and exercise and stable metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes that has been treated with lifestyle modification and a stable dose of metformin ≥1000 mg/day (or maximum tolerated dose) for at least 3 months at the time of Screening
* Screening HbA1c 7.0-10.5%
* Male or female, age 18-75 years
* Screening BMI 24.5 - 40 kg/m2
* Either surgically sterile, abstinent, or willing to use a highly effective method of contraception for the entirety of the study, and not be pregnant or lactating if a woman of child-bearing potential

Exclusion Criteria:

* Has received within the preceding 3 months prior to Screening, another approved or investigational oral or injectable antidiabetic medication (including, but not limited to sulfonylureas, dipeptidyl peptidase-4 inhibitor [DPP-4i], sodium-glucose cotransport 2 inhibitors, alphaglucosidase inhibitors, meglitinides, thiazolidinediones) or insulin in addition to metformin therapy
* Has active GI disease including acute or chronic pancreatitis, severe gastroparesis or chronic malabsorption, inflammatory bowel disease, symptomatic gallbladder or biliary disease, known unstable liver disease, a diagnosis of fibrotic nonalcoholic steatohepatitis (NASH), Gilbert's syndrome, or obvious clinical signs or symptoms of liver disease including chronic active hepatitis B or C, or primary biliary cirrhosis, or elevated alanine aminotransferase (ALT) levels at Screening
* Has any history of myocardial infarction (MI), unstable angina, coronary artery bypass graft, percutaneous coronary therapeutic intervention, transient ischemic attack, stroke, or decompensated congestive heart failure within previous 6 months prior to Screening
* Has an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2
* Has active proliferative diabetic retinopathy or macular edema
* Has a known self or family history (first-degree relative) of multiple endocrine neoplasia type 2A or type 2B, thyroid C-cell hyperplasia, or medullary thyroid cancer
* Has an active or untreated malignancy or has been in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for <5 years prior to screening
* Has evidence of human immunodeficiency virus (HIV) and/or positive HIV antibodies historically or at screening
* Has had a significant change in weight, defined as a gain or loss of at least 5% body weight in the 3 months prior to screening
* Has been treated or plan to be treated with drugs or devices or surgery that promote weight loss within 3 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to end of treatment in the modified intent-to-treat population | up to 16 weeks

SECONDARY OUTCOMES:
Change in fasting plasma glucose from baseline to end of treatment in the modified intent-to-treat population | up to 16 weeks
Change in mean body weight (absolute and %) from baseline to end of treatment in the modified intent-to-treat population | up to 16 weeks
Change in body mass index from baseline to end of treatment in the modified intent-to-treat population | up to 16 weeks
Change in waist circumference from baseline to end of treatment in the modified intent-to-treat population | up to 16 weeks
Change in mean blood lipids including triglycerides (TG), high-density lipoprotein (HDL), and low-density lipoprotein (LDL) from baseline to end of treatment in the modified intent-to-treat population | up to 16 weeks
Percentages of patients achieving HbA1c <6.0%, <6.5%, and/or <7.0% | up to 16 weeks
Percentages of patients achieving ≥5% and/or ≥10% greater body weight loss | up to 16 weeks
Incidence of treatment-emergent adverse events (TEAE)s, serious adverse events (SAE)s, deaths, and adverse events (AE)s leading to study discontinuation | up to 16 weeks
Vital signs - Systolic blood pressure (mmHg) absolute change from baseline | up to 16 weeks
Vital signs - Diastolic blood pressure (mmHg) absolute change from baseline | up to 16 weeks
Vital signs - Heart rate (beats/minute) absolute change from baseline | up to 16 weeks
Vital signs - Body weight (kg) absolute and percent change from baseline | up to 16 weeks
Safety clinical laboratories - complete blood count absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum sodium absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum potassium absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum total bilirubin absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum direct bilirubin absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum alkaline phosphatase absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum alanine aminotransferase absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum aspartate aminotransferase absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum blood urea nitrogen absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum creatinine absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum uric acid absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum calcium absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum lipase absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum amylase absolute change from baseline | up to 16 weeks
Safety clinical laboratories - eGFR (calculated) absolute change from baseline | up to 16 weeks
Safety clinical laboratories - fasting serum glucose absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum albumin absolute change from baseline | up to 16 weeks
Safety clinical laboratories - serum total protein absolute change from baseline | up to 16 weeks
Safety clinical laboratories - fasting serum total cholesterol absolute change from baseline | up to 16 weeks
Safety clinical laboratories - fasting serum triglycerides absolute and percent change from baseline | up to 16 weeks
Safety clinical laboratories - fasting serum HDL-C absolute and percent change from baseline | up to 16 weeks
Safety clinical laboratories - fasting serum LDL-C absolute and percent change from baseline | up to 16 weeks
Safety clinical laboratories - serum calcitonin absolute change from screening | up to 16 weeks
ECG interval change from baseline absolute and categorical outliers >450ms | up to 16 weeks
Proportion of patients who report AEs of Special Interest (AESI) including GI intolerability, hypoglycemia, drug hypersensitivity reactions, acute pancreatitis, thyroid C-cell hyperplasia and C-cell neoplasms, and cardiovascular (CV) events | up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Axon Clinical Research, Doral, Florida, United States